CLINICAL TRIAL: NCT04950439
Title: Pyrophosphate: a New Biomarker to Predict Arterial Calcification in Chronic Kidney Disease
Brief Title: Pyrophosphate and Arterial Calcification in Chronic Kidney Disease
Acronym: Predical
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-API-02
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myocardial CT (Other): The investigator will collect the usual clinical history and data. Risk factors and cardiovascular events are identified. A blood sample dedicated to the study and necessary for routine care is taken. The pulse wave velocity and systolic pressure index are measured. A myocardial CT scan coupled with a computed tomography is performed. The patient collects stools at his home, simply conditions them and sends them by mail to the centre, which stores them.
  Interventions: Other: Collect blood sample

INTERVENTIONS:
Other: Collect blood sample — A blood sample dedicated to the study and necessary for routine care is taken. The pulse wave velocity and systolic pressure index are measured. A myocardial CT scan coupled with a computed tomography is performed. The patient collects stools at his home, simply conditions them and sends them by mail to the centre, which stores them.

SUMMARY:
Arterial calcifications start at early stages of chronic kidney disease (CKD) and are associated to cardiovascular mortality. Pyrophosphate (PPi) is an endogenous compound, which stops the mineralization process in bones and is expected to act at ectopic sites. In uremic rats, low PPi plasma levels are associated with high calcium content in the aorta and peritoneal administration of PPi blocks this process. People on maintenance dialysis or kidney transplant recipients have low plasma levels of PPi and show high scores of arterial calcification. The purpose is to determine the role of low PPi in the development of arterial calcifications in patients with CKD stage 3 or 4. To that aim, 252 patients with eGFR between 59 et 20 ml/min/1,73 m2 will be recruited and will be examined at baseline and three years later.

ELIGIBILITY:
Inclusion Criteria:

* eGFR between 59 et 20 ml/min/1,73 m2 twice at three month interval

Exclusion Criteria:

1. kidney transplantation
2. acute inflammatory disease or active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of PPI | 3 years
  To show that low plasma levels of PPi at baseline is associated with a high progression of arterial calcification at three years after adjustment for confounding variables

CONTACTS AND LOCATIONS:
Overall Officials: Favre Guillaume, PhD, Principal Investigator — CHU de Nice, Service de Néphrologie
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided